CLINICAL TRIAL: NCT01927263
Title: A Phase 3 Clinical Study of NI-071 in Patients With Rheumatoid Arthritis -A Double-blind, Active Drug-controlled Study and Long-term Study-
Brief Title: A Phase 3 Study of NI-071 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nichi-Iko Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI071F1(EFC13464)
Record Dates: First submitted 2013-08-09; First posted 2013-08-22 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NI-071 (Experimental)
  Interventions: Biological: NI-071
- Infliximab (Active Comparator)
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: NI-071 — 100mg/vial
  Arms: NI-071
Biological: Infliximab — 100mg/vial
  Other Names: Remicade
  Arms: Infliximab

SUMMARY:
The purpose of this study is to investigate similarity between NI-071 and infliximab(the comparator) in terms of efficacy in patients with Rheumatoid Arthritis not adequately responding to Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of RA as defined by the American College Rheumatology (ACR) and European League Against Rheumatism (EULAR) criteria (ACR/EULAR 2010)
2. Patients who received MTX treatment (6- 16mg/week) for 2 weeks for at least 12 weeks prior to the screening visit

Exclusion Criteria:

1. Patients with a following past History or concomitant diseases

   * Other Connective tissue disorders which may interfere the efficacy assessment
   * Chronic or recurrent infectious disease
   * Demyelinating disease
   * Congestive heart failure
   * lymphoproliferative disorder or myelodysplastic syndrome
   * Malignancy
   * Interstitial lung disease
2. Patients with active or latent tuberculosis or history of tuberculosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Efficacy : Changes in DAS28-ESR | week 0 to week 14

SECONDARY OUTCOMES:
Efficacy : Changes in DAS28 | week 0 to week 54
Efficacy : Changes in ACR20, 50, 70 | week 0 to week 54
Efficacy : Changes in ACR core-set | week 0 to week 54
Safety : Long term safety (Adverse Events, Immunogenicity, etc.) | to 54 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NichiIko Investigational Site, Sendai, Japan